CLINICAL TRIAL: NCT05281575
Title: Evaluation of the Psychosocial Impacts of Baby Friendly Spaces for Rohingya Refugee Mothers Living in Cox's Bazar, Bangladesh.
Brief Title: Evaluation of Baby Friendly Spaces in Cox's Bazar, Bangladesh.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Action Contre la Faim (Other)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other); University of Virginia (Other); University Research Co, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FRGB2B-FR27; FY21-A01-6024 (Other Grant/Funding Number: University Research Co., LLC)
Record Dates: First submitted 2022-02-09; First posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Psychosocial Functioning; Psychological Distress
Keywords: Psychosocial intervention; Refugees; Maternal health; Bangladesh

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The co-PIs are masked, as are data analysts. The participants have not been told what arm of the trial they are in, and outcome assessors assigned to integrated nutrition centers have not been told if that center was re-trained or not, though it is conceivable that they could deduce this information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual BFS (TAU BFS) (Active Comparator): Continuation of existing Baby Friendly Spaces program activities in integrated nutrition centers, which are not manualized and without re-training have naturally drifted in fidelity to the intervention and supervision approach due to time since initial training.
  Interventions: Behavioral: Baby Friendly Spaces (BFS)
- Enhanced BFS (Experimental): The implementation-enhanced BFS intervention includes re-training using newly developed training materials that focus on building core therapeutic engagement skills. Ongoing supports include brief guidance sheets for each of the most commonly delivered BFS activities, as well as newly established group supervision focused on BFS, discussion facilitation, activities and self-care.
  Interventions: Behavioral: Baby Friendly Spaces (BFS)

INTERVENTIONS:
Behavioral: Baby Friendly Spaces (BFS) — Designed to meet the unique needs of populations living in humanitarian contexts, BFS focus on two domains: psychosocial support that targets maternal wellbeing and childcare practices that target caregiver functioning to also address child wellbeing and development. In so doing, BFS strengthens mothers' internal resources and skills in caring for their children both in quantity (time spent caring for the child) and quality (responsiveness), to positively impact the health status and wellbeing of their children. In BFS, the following activities are delivered by trained psychosocial workers: counselling for infant and young child feeding practices; hygiene education and promotion; mother-child bonding activities that provide psychosocial stimulation essential for children at risk of, or experiencing, malnutrition; and provision of maternal psychosocial support (i.e. psychoeducation, stress management).

SUMMARY:
The overarching goal of this study is to evaluate the effectiveness and implementation of the Baby Friendly Spaces (BFS) program for improvement of maternal psychosocial wellbeing among Rohingya refugee mothers and their malnourished infants and young children in Cox's Bazar, Bangladesh. The purpose of the BFS program is to provide convenient, accessible psychosocial support to mothers in order to facilitate their ability to care for their children. BFS activities include: counselling for infant and young child feeding practices, hygiene education and promotion, group discussions on parenting skills, mother-child bonding activities and maternal psychosocial support. In Cox's Bazar, the BFS program is not currently standardized as intended. In this study, integrated nutrition centers that offer the BFS program are being paired and randomized to receive re-training in a standardized and implementation-enhanced version of BFS (enhanced-BFS) or to continue BFS services as usual (TAU-BFS). Primary (symptoms of psychological distress and functional impairment) and secondary (subjective psychosocial wellbeing and coping) outcomes will be assessed immediately post intervention (8 weeks after initial baseline assessment) via interviewer-administered surveys. The central hypothesis is that mothers attending enhanced-BFS services will experience greater improvement in all psychosocial well-being indicators relative to mothers in the standard, treatment-as-usual centers.

DETAILED DESCRIPTION:
Action contre la Faim (ACF) currently provides psychosocial support services to Rohingya mothers of malnourished children who are receiving nutrition support at Integrated Nutrition Centers (INCs) within refugee camps in Cox's Bazar, Bangladesh. At the INCs, the Baby Friendly Spaces (BFS) program is offered as a part of ACF's psychosocial and care practices support strategy. The BFS program is a holistic psychosocial support program designed to enhance mothers' wellbeing in order to buffer against the deleterious health and developmental impacts of conflict and disaster on children. BFS is designed to be flexible to meet the unique needs of different conflict-affected populations using a community-based approach, but always focuses on two domains: psychosocial support that targets maternal wellbeing and childcare practices that target caregiver functioning to also address child wellbeing and development. In so doing, BFS strengthens mothers' internal resources and skills in caring for their children to positively impact the nutritional status and wellbeing of their children during humanitarian emergencies. The purpose of this study is to evaluate the effectiveness of the BFS program for improving the psychosocial wellbeing of Rohingya refugee mothers of young (ages 0-2) children experiencing malnutrition in Cox's Bazar, Bangladesh.

As they are currently functioning, BFS activities in Cox's Bazar are not standardized as intended. Thus, this study will use a pre-post, paired randomized study design to compare two conditions being delivered within Integrated Nutrition Centres (INCs) in Cox's Bazar-based refugee camps: 1) treatment-as-usual BFS mental health and psychosocial support prevention and promotion activities (TAU BFS) as they are currently being offered; and 2) implementation-enhanced BFS activities (enhanced-BFS) that includes intervention standardization, re-training, and implementation supports. The primary outcomes being evaluated are symptoms of psychological distress and functional impairment, and secondary outcomes include subjective maternal wellbeing and coping skills. Although a randomized controlled trial (RCT) comparing BFS against a non-active control condition would provide the clearest evidence, such a design is not feasible in this context because the services are already being offered as a part of existing programming, and removal of any existing supports would be unethical. As such, the proposed study design uses current BFS practices occurring in Integrated Nutrition Centers (INCs) that have not been manipulated as part of the research (treatment as usual). These services are not manualized and have been affected by natural drifts in fidelity over time since initial training. In the intervention condition, psychosocial workers and psychologists at select INCs will be re-trained in a manualized version of the BFS program, and will continue to receive additional implementation support during the study through newly established supervision structures (enhanced-BFS).

As the experimental manipulation is occurring at the INC-level, INCs were paired by overseeing psychologist (as in some cases one psychologist oversees two sites) and randomize within the pair to intervention (BFS-enhanced) or treatment as usual control (BFS TAU). In addition to incorporating site matching in the design phase to help try to minimize bias in group comparisons while assessing the intervention as implemented in the real world, propensity score adjustments in the analysis approach will be leveraged. After completing the BFS intake, eligible and interested mothers are referred to a data collector to obtain informed consent and administer a baseline interview. Mothers can then participate in BFS to whatever extent they choose. The same data collector will follow up with each mother 8-10 weeks later to complete a follow-up interview. Because of logistical constraints, each INC has been assigned a single data collector to carry out study activities at that site. All sites will also record detailed information (as part of regular program monitoring) about activities delivered and received by women enrolled in BFS at the INCs. Two trained observers will rotate through the INCs to record fidelity data. This real-world comparison of an intervention implemented "as is" versus an enhanced program implemented with effort towards greater standardization and fidelity will provide insight about effectiveness of the program model and structures and resources that need to be in place to effectively implement the program.

ELIGIBILITY:
Inclusion Criteria:

* Adult (aged 18 or older) Rohingya women enrolling for the first time in BFS services at a participating integrated nutrition center (INC)
* The mother of a child under age 2 who is identified as suffering from moderate or severe acute malnutrition without complication by ACF
* Able to speak and understand Chittagonian dialect of Bangla

Exclusion Criteria:

* Target child has a severe developmental disability or is severely malnourished with complications
* Maternal cognitive impairment or psychosis that would preclude participation in program activities
* Referred per standard program practice to more specialized mental health or protection services outside of Action Contre la Faim (ACF)
* Planning to leave the area in the next 2 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2021-11-28 (Actual); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Symptoms of psychological distress by a combined IDSS and K-6 | Baseline (pre), 8 weeks (post)
  Change in mean score on an adapted psychological distress scale comprised of items from the Myanmar-wide version of the International Depression Symptom Scale (IDSS) questionnaire as well as the Kessler-6. Together, these items assess common indicators of psychological distress including symptoms of depression, anxiety, and somatic complaints. Prior to generating scale scores, baseline data will be used to examine the scale's psychometric properties including factor structure and internal consistency, and will remove any problematic items. Higher scores indicate greater symptom severity.
Functional Impairment by the WHO Disability Assessment Schedule 2.0 (WHODAS) | Baseline (pre), 8 weeks (post)
  Change in mean score of the WHODAS 2.0 questionnaire assessing six domains of functioning: cognition, mobility, self-care, getting along/social interactions, life activities, and participation. Each item is coded either "none", "mild", "moderate", "severe" and "extreme". The total score ranges between 0 and 60. Higher scores indicate greater disability severity.

SECONDARY OUTCOMES:
Subjective Well-Being by the Personal Well-being Index-Adult (PWI-A) | Baseline (pre), 8 weeks (post)
  The Personal Well-being Index-Adult (PWI-A) assesses satisfaction with specific life domains, e.g., health, safety, personal relationships etc. Each item is rated on a likert scale from 0 (no satisfaction at all) to 10 (very satisfied). Change scores will be calculated for both overall wellbeing as well as domain-specific wellbeing. Scored between 0- 100. Higher scores indicate greater satisfaction.
Coping styles by the Brief COPE | Baseline (pre), 8 weeks (post)
  Coping styles will be assessed using an adapted version of the Brief COPE (26 items) that includes addition of items previously generated from qualitative study in this population as well as removal of items identified during pre-testing to be redundant, irrelevant, or difficult-to-understand. the scale defines the primary copng style among three coping styles. Scored between 0-78. The higher score indicate higher engagement in a coping style.

OTHER OUTCOMES:
Qualify of caregiving practices | Baseline (pre), 8 weeks (post)
  Change scores using a brief, program-developed questionnaire that assesses care practices (i.e. responsive feeding and child psychosocial stimulation) and feelings towards the child. Scored between 0-21.
Implementation outcomes | 8 week follow-up
  Between-group difference in mean scores on implementation domains assessed using the Mental Health Implementation Science Tools (mhIST) consumer and provider versions. These have been validated across multiple mental health and psychosocial support studies and assess adoption, acceptability, appropriateness, and feasibility of the intervention.
Child growth and development by the WHO Gross motor development milestones | 8 week follow-up
  Five milestones are considered to be universal and fundamental to the acquisition of self-sufficient locomotion skills. The child's performance (last milestone reached) is recorded based on the mother's observation. The scored ranges between 0-5 and ages of achievement outside the windows of reference is indicative of a motor delay

CONTACTS AND LOCATIONS:
Overall Officials: Karine LE ROCH, PhD, Principal Investigator — Action Contre la Faim; Sarah MURRAY, PhD, Principal Investigator — Jonhs Hopkins University; Amanda NGUYEN, PhD, Principal Investigator — University of Virginia
Locations (1):
- Action Against Hunger, Cox’s Bāzār, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
De-identified quantitative survey data will be shared in USAID's Developmental Data Library
Supporting Information: Analytic Code
Time Frame: Beginning six months after publication of summary data, to remain available until USAID determines removal from Developmental Data Library.